CLINICAL TRIAL: NCT06427356
Title: PREVAIL: Efficacy of a Veterans Healthcare Administration (VHA) Whole Health Interdisciplinary Pain Clinic
Brief Title: PREVAIL Interdisciplinary Track: A Pragmatic Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salem Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Durham VA Health Care System (U.S. Federal Agency); VISN 6 MIRECC (Unknown); Bedford VA Health Care System (Unknown); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC 0004
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
Keywords: Whole health; rural health; Interdisciplinary team
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary Team (Experimental): Participants complete surveys, meet with five pain specialists to develop individualized treatment plans based on whole health, receive monthly coaching calls for five months, then meet with the pain specialists once more for a 6-month follow-up appointment and complete surveys.
  Interventions: Behavioral: PREVAIL Interdisciplinary Team
- Waitlist Control (No Intervention): Participants complete surveys but do not engage with the pain specialists for 6 months.

INTERVENTIONS:
Behavioral: PREVAIL Interdisciplinary Team — Patient meets simultaneously with an interdisciplinary team (IDT) five pain specialists and develops an individualized treatment plan based on Whole Health. Participants receive five months of coaching calls then return six months later for a follow-up visit with the IDT.
  Arms: Interdisciplinary Team

SUMMARY:
The goal of this clinical trial is to [primary purpose learn if a team that involves five types of pain specialists (interventional pain, psychology, pharmacy, nutrition, physical therapy) can treat chronic pain in Veterans. The main questions it aims to answer are:

* Do patients report less pain after six months in the program?
* Do patients report that pain gets in the way of their life less after six months in the program? The researchers will compare participants who participate in the program to those that wait for six months before participating in the program.

Participants will

* Meet with the team of pain specialists to develop a plan to treat their pain
* Receive calls from a coach once per month
* Return to meet with the team of pain specialists for a six-month follow-up appointment
* Fill out surveys

ELIGIBILITY:
Inclusion Criteria:

* Veteran receiving care at the Salem VA Health Care System (Salem VAHCS) per electronic medical record (EMR)
* Patient participating in PREVAIL Interdisciplinary Team Track per EMR
* Chronic Pain Diagnosis: Defined as pain lasting more than three months per EMR

Exclusion Criteria:

* Diagnosis of Mild Neurocognitive Disorder or Major Neurocognitive Disorder based on Diagnostic Statistical Manual of Mental Disorders, 5th edition, Text Revision (DSM-5-TR) per EMR
* Veteran has a current acute physical injury that would artificially elevate pain scores during study period per EMR
* Veteran intends to have a pain-related surgery during the study period per EMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Baseline, 6-months
  A 9-item scale used to quantify an individual's pain experience (0-10) with higher scores suggesting worse pain severity and pain interference.

SECONDARY OUTCOMES:
Short Form-36 Item (SF-36) | Baseline, 6-months
  A 36-item scale to assess quality of life, including any impact of health problems on completing activities, as well as energy and emotions, with lower scores indicating a higher impact of health problems.
Insomnia Severity Index | Baseline, 6-months
  A 7-item scale that assesses sleep disturbances, with higher scores reflecting more sleep difficulty.
Pain Self-Efficacy Questionnaire | Baseline, 6-months
  A 10-item scale used to determine how confident an individual is in accomplishing tasks despite the pain (0=not at all confident and 6= completely confident) with higher scores denoting higher levels of pain self-efficacy.
University of Washington- Concerns about Pain Scale 24-item | Baseline, 6-months
  A 24-item scale used to assess one's perception of their pain experience (1= never, 5= always), with higher scores indicating higher levels of pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Rena E Courtney, PhD, Principal Investigator — Salem VA Health Care System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Courtney RE, Schadegg MJ. Chronic, Noncancer Pain Care in the Veterans Administration: Current Trends and Future Directions. Anesthesiol Clin. 2023 Jun;41(2):519-529. doi: 10.1016/j.anclin.2023.02.004. Epub 2023 Mar 15. PMID 37245954
- [Background] Darnall BD, Edwards KA, Courtney RE, Ziadni MS, Simons LE, Harrison LE. Innovative treatment formats, technologies, and clinician trainings that improve access to behavioral pain treatment for youth and adults. Front Pain Res (Lausanne). 2023 Jul 20;4:1223172. doi: 10.3389/fpain.2023.1223172. eCollection 2023. PMID 37547824
- [Background] Courtney RE, Schadegg MJ, Bolton R, Smith S, Harden SM. Using a Whole Health Approach to Build Biopsychosocial-Spiritual Personal Health Plans for Veterans with Chronic Pain. Pain Manag Nurs. 2024 Feb;25(1):69-74. doi: 10.1016/j.pmn.2023.09.010. Epub 2023 Oct 13. PMID 37839983